CLINICAL TRIAL: NCT04625621
Title: Breast Reconstruction by Exclusive Lipomodulin : Feasibility, Evaluation of the Aesthetic Result and Quality of Life
Acronym: EXCLUFAT
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2020-22
Record Dates: First submitted 2020-10-07; First posted 2020-11-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the leading female cancer in metropolitan France in terms of incidence and death. Among the therapeutic arsenal for the treatment of these cancers, surgery plays a very important role and even if a conservative treatment is possible in the majority of cases, there is still an indication for mastectomy in about 30% of cases.

Currently, only 30% of women who have undergone a mastectomy choose reconstruction.

The primary objective of breast reconstruction from a surgical point of view is to leave as few aesthetic and functional after-effects as possible while meeting the personal wishes of each woman according to her morphological, tissue and vascular characteristics.

There are currently 2 major surgical procedures for breast reconstruction: breast implant reconstructions and autologous reconstructions.

Breast reconstruction by prosthesis is the simplest and most widely used technique but, the controversies concerning implants with the PIP breast prostheses scandal in 2010 and more recently the anaplastic lymphoma scandal have tarnished the image of this type of reconstruction.

Alternatives to breast implants have been developed: autologous reconstructions using first pedicled tissue flaps, then free flaps, techniques that allow a more natural, more satisfactory aesthetic result with an evolution that follows the patient's own morphology but requiring specific training in microsurgery and not without postoperative complications.

Since 1999, the investigators have witnessed the evolution of another autologous technique, that of lipomodulin. Initially used to improve the results of reconstructions and the aesthetic sequelae of conservative treatments, it is now used as an exclusive reconstruction technique. Easily reproducible and offering several advantages, reconstruction by exclusive lipomodulin is increasingly appreciated by patients.

However, this increasingly practiced technique presents specific problems and this is what the investigators want to evaluate in this study.

The main objective of this study is to evaluate the practices within our establishment regarding breast reconstruction by exclusive lipomodulin in terms of feasibility. The secondary objectives are the evaluation of the cosmetic result and the quality of life of these patients after this type of reconstruction.

DETAILED DESCRIPTION:
This is an observational, monocentric study using retrospective health data (2012-2020) combined with quality of life questionnaires.

The list of patients meeting the inclusion criteria will be collected using the Medical Information Department. Based on a screening of aggregate data from the center, the sample size is approximately 150 patients.

The questionnaires will be mailed to patients during a follow-up site visit:

* The WHOQOL-BRIEF
* The EXCLUFAT questionnaire
* The questionnaire to be completed by a third party. A phone call will be made to explain the principle of the study and answer any questions they may have.

The returned questionnaires will be analyzed. Other necessary data will be collected in the patients' computer files.

There is no provision for patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Patient who benefited from immediate or delayed breast reconstruction by exclusive lipomodulin completed between 01/01/2012 and 07/31/2020.
3. Agreeing to answer the questionnaire

Exclusion Criteria:

1. Association with another prosthetic or autologous reconstruction technique planned at the beginning of the reconstruction procedure.
2. Deceased patient
3. Patient under guardianship or curators
4. Patient opposed to the use of her data for research

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient treated by mastectomy for breast cancer having completed an exclusive lipomodeling reconstruction course (immediate or delayed reconstruction) at the ICO - Saint Herblain site between January 2012 and July 2020.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of the exclusive lipomodulin technique in breast reconstruction: Failure rate of the technique | 18 months
  Failure rate of the technique

SECONDARY OUTCOMES:
Evaluate the aesthetic result | 18 months
  Scale of evaluation of the aesthetic result by a third party (specific scale with 4 question/scale form 1 to 10).
Evaluate patient satisfaction: BREAST-Q | 6 months
  BREAST-Q (Reported Outcome Assessment following Reconstructive Breast Surgery in 31 questions including 10 scale from 1 to 10)
Assessing patient quality of life: WHOQOL BREF | 6 months
  World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall QOL and general health.

CONTACTS AND LOCATIONS:
Overall Officials: BRILLAUD-MEFLAH Victoire, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancerologie de L'Ouest, Saint-Herblain, France